CLINICAL TRIAL: NCT06677034
Title: Effect of Mobile Game-Based Exercise Training on Functional Performance, Brain-Derived Neurotrophic Factor, Executive Functions and Sleep Quality in Children with Epilepsy
Brief Title: Effects of Exercise on Functional Performance, BDNF, Executive Functions and Sleep Quality in Children with Epilepsy
Acronym: BDNF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Filiz Özdemir, ASSOC. PROF. DR., Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-KAEK-08
Record Dates: First submitted 2024-10-25; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Epilepsy
Keywords: epilepsy; BDNF; child; functional performance; sleep quality; executive functions
MeSH Terms: conditions — Epilepsy; Sleep Initiation and Maintenance Disorders | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (No Intervention)
- intervention (Experimental): Consent will be obtained from the volunteer children and parents and a WhatsApp group will be established. Parents will be asked to fill out sociodemographic forms about themselves and the child. Students whose parents have given their consent will be included in the study and a mobile game-based exercise program will be started. Each online animated game-based exercise program will be supervised by a researcher physiotherapist. Game-based exercise program sessions with animated characters will be planned for 12 weeks/3 days a week/30 minutes. Fatigue perceptions will be assessed with the Modified Borg Scale after each exercise. Children who show any symptoms will take a break from the session. The first assessment will be made before the sessions start and the final assessment will be made after the 12-week exercise program.
  Game-based exercise program content:
  Warm-up Exercise Program Warm-up exercise training; fun and interesting animated game-based exercise that will allow the hea
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Mobile Game-Based Exercise Training
  Arms: intervention

SUMMARY:
According to the definition of the International League for the Control of Epilepsy, a seizure is the emergence of temporary symptoms and/or findings as a result of abnormal, excessive and simultaneous stimulation of neurons in the brain. Epilepsy is a state of being prone to recurrent seizures; epilepsy is at least two seizures that occur without a cause that can be shown at the time and recur within more than 24 hours. Approximately one in 150 children is diagnosed with epilepsy in the first 10 years of their life, and the highest incidence rate is seen in infancy. A study conducted on individuals with epilepsy has indicated that exercise can create positive neuronal changes and reduce damage. In this context, 50 children with epilepsy between the ages of 6 and 10 who are being followed up at the Department of Child Neurology at Malatya Education and Research Hospital will be selected for the study and will be divided into experimental and control groups. In the randomized controlled study, the experimental group will be given mobile game-based exercise training, while the control group will not receive any intervention. Functional performance, BDNF, executive functions and sleep quality will be assessed in both groups at the beginning of the exercise and after the completion of the 12-week mobile game-based exercise intervention. Functional performance assessment will be performed using the timed up and walk test and the timed stair ascent and descent test. BDNF levels will be determined from the blood. The BRIEF-Parent Form will be used to assess executive functions. The Childhood Sleep Disorder Scale will be used for sleep quality. The aim of the study is to evaluate the effects of mobile game-based exercise training on functional performance, brain-derived neurotrophic factor, executive functions and sleep quality in children with epilepsy.

DETAILED DESCRIPTION:
According to the definition of the International League Against Epilepsy, a seizure is the emergence of temporary signs and/or symptoms as a result of abnormal, excessive and simultaneous stimulation of neurons in the brain. Epilepsy is a state of being prone to recurrent seizures; epilepsy is at least two seizures that occur without a cause that can be demonstrated at the time and recur within more than 24 hours. Approximately one in 150 children is diagnosed with epilepsy in the first 10 years of their life, with the highest incidence rate seen in infancy. Recent studies conducted in different populations in Turkey have indicated that the incidence of epilepsy in children and adolescents is between 20 per 100,000 and 124 per 100,000. Families of children with epilepsy report high levels of stress (45%), depression (46%) and anxiety (56%). The concept of gamification is based on the application of "game design elements in a non-game context" to motivate participation. Many studies have reported the positive effects of game-based education in children. Through play, the child's psychomotor skills, strength, reaction and attention are increased, control of large and small muscles is taken under control and balance, flexibility and agility are provided in movements.

Studies on the subject show that exercise can create positive neuronal changes in individuals with epilepsy and reduce damage. Regular exercise is associated with changes in neurotransmitter levels, glial cell volume, expression of endogenous neurotrophic factors and increased neurogenesis. Considering these neurobiological effects of exercise, physical activity has been shown to have beneficial effects on neurodegenerative diseases.

Functional performance refers to certain activities and behaviors that individuals can perform at a certain level in daily life. It is known that functional performance is affected in children with epilepsy. When the literature is examined, it has been seen that children and adolescents with epilepsy but without additional disabilities have surprisingly high motor problems, especially in the areas of reaction speed, balance and coordination.

Brain-derived neurotrophic factor (BDNF) belongs to the neurotrophin family, which are growth factors that have trophic effects on neurons. BDNF is the most widely distributed neurotrophin in the central nervous system and is highly expressed in the prefrontal cortex and hippocampus. It is generally accepted that BDNF plays a role in synaptic plasticity by regulating presynaptic and postsynaptic transmission. There are studies showing that BDNF levels are altered in individuals with epilepsy.

Sleep disorders are more common in children with epilepsy than in the general population. Due to the bidirectional relationship between epilepsy and sleep disorders, it is extremely important to evaluate sleep disorders in individuals with epilepsy. At the same time, behavioral changes, cognitive problems, and learning difficulties (mostly attention problems and hyperactivity) are more common in children with epilepsy, 24-66% more than in the general population; these changes are strongly associated with insomnia or excessive sleepiness.

Epilepsy in childhood is characterized as a chronic medical disease with a characteristic behavioral and cognitive phenotype that includes impaired executive functions and attention-related deficits. Studies have shown that executive functions are affected in children with epilepsy. In the literature, the sample group of studies on the effects of exercise in epilepsy is usually adults. In this case, data on the effects of exercise in children with epilepsy are quite limited. This study will evaluate the effects of exercise training on functional performance, brain-derived neurotrophic factor, executive functions and sleep quality in children with epilepsy and will provide data and contributions to fill this gap in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with G40 (epilepsy) between the ages of 6-10
* Epileptic seizures under control
* No additional neuromuscular, psychiatric, orthopedic, cognitive function, etc. problems
* Presence of a device that will provide regular mobile application access
* Ability to use the mobile application
* Volunteering of the family and child to participate in the study

Exclusion Criteria:

* Having a condition that prevents performing exercises and tests

  * Having a psychosocial problem that prevents adaptation to the study
  * Having an auditory, visual, etc. disability
  * Having a seizure in the last 6 months
  * Having a regular exercise or sports habit
  * Other diseases that will cause difficulty in perceiving the instructions given to the person
  * Patients who do not give informed consen

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-12-23 (Estimated)

PRIMARY OUTCOMES:
bdnf | 3 month
  The change in BDNF levels in the blood will be checked before and after 3 months of exercise.
functional performance | 3 month
  will be evaluated with timed up and walk test .Changes will be examined before and after 3 months of exerciseTime
functional performance | 3 month
  will be evaluated stair climbing test . Changes will be examined before and after 3 months of exerciseTime
sleep quality | 3 month
  Will be evaluated with Children's Sleep Disorder Scale.On a five-point Likert-type scale, 1 corresponds to 'never', while 5 corresponds to 'always (daily)'. Higher scores indicate more acute sleep disturbances
executive function | 3 month
  will be evaluated with the brief parent form

IPD SHARING:
Plan to Share IPD: No